CLINICAL TRIAL: NCT02748655
Title: Alkaline Ionized Water: Sports Recovery and Inflammation Management
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Principal Investigator, Gitte Jensen, Ph.D., Research Director, Natural Immune Systems Inc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NIS119004
Record Dates: First submitted 2016-03-11; First posted 2016-04-22 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Sports Recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tap water (Placebo Comparator): Oral consumption of tap water
  Interventions: Other: Tap water
- Alkaline ionized water (Active Comparator): Oral consumption of alkaline ionized water
  Interventions: Other: Alkaline ionized water

INTERVENTIONS:
Other: Alkaline ionized water
  Arms: Alkaline ionized water
Other: Tap water
  Arms: Tap water

SUMMARY:
The purpose of this study is to determine whether consumption of alkaline ionized water is effective for accelerating sports recovery.

DETAILED DESCRIPTION:
Alkaline ionized water versus tap water is consumed for one week prior to an exercise challenge, using a cross-over study design.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age 25-40 years (inclusive)
* Body mass index (BMI) between 19.0 and 29.9 kg/m2 (inclusive)
* Not regularly exercising or participating in team sports.

Exclusion Criteria:

* Bariatric surgery
* Diagnosed and medicated for diabetes
* Known serious chronic health condition
* Serious active illness within past 12 months
* Major surgery during past 8 weeks
* Alcohol consumption of more than four standard units/day (for example more than four regular 12-oz beers (5% alcohol), four small 5-oz glasses of wine (12% alcohol), or four 1.5 oz shots of 80-proof spirits) (or more than 28 per week);
* Regular use of marijuana products for the past three months
* Regular consumption of energy drinks
* Diagnosed with any blood clotting disorder or taking clotting factor concentrates.
* Taking any blood thinners or anticoagulants
* Taking anti-inflammatory medications on a daily basis (81 mg aspirin is acceptable)
* Diagnosed with high blood pressure or taking blood pressure medication
* Use of performance enhancing drugs within the last three months
* Having consumed prednisone (or related steroid medication) or received a prednisone injection within the last six months

Ages: 25 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Plasma lactate levels | One hour
  Plasma lactate levels will be measured five times (at 15-minute intervals) within one hour after performing high intensity interval training exercise.

SECONDARY OUTCOMES:
Complete Blood Count | One hour
  Complete blood count with differential will be performed immediately after, and at 1 hour after, performing high intensity interval training exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte S Jensen, PhD, Principal Investigator — Natural Immune Systems Inc
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No